CLINICAL TRIAL: NCT00577278
Title: A Phase II Study of Allogeneic Hematopoietic Stem Cell Transplant for B-Cell Non-Hodgkin Lymphoma Using Zevalin, Fludarabine and Melphalan
Brief Title: A Phase II Study of Allo-HCT for B-Cell NHL Using Zevalin, Fludarabine and Melphalan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05149; P01CA030206 (NIH); CHNMC-05149; CDR0000579136 (Registry Identifier: NCI PDQ); NCI-2010-01230 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Results first posted 2022-12-23 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma
Keywords: graft versus host disease; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; recurrent adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; Waldenstrom macroglobulinemia; contiguous stage II marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; recurrent adult diffuse mixed cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — Rituximab; fludarabine phosphate; Melphalan; Sirolimus; Tacrolimus; Indium; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemo, monoclonal antibody therapy, transplant) (Experimental): REDUCED-INTENSITY CONDITIONING: Patients receive rituximab IV followed by indium In-111 ibritumomab tiuxetan IV over 10 minutes on day -21 and rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day -14. Patients also receive fludarabine phosphate IV on days -9 to -5 and melphalan IV on day -4. STEM CELL TRANSPLANTATION: Patients undergo APBSCT on day 0. GVHD PROPHYLAXIS: Patients receive tacrolimus IV or PO and sirolimus PO beginning on day -3 and continuing for up to 6 months with taper.
  Interventions: Biological: rituximab; Drug: fludarabine phosphate; Drug: melphalan; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Radiation: indium In 111 ibritumomab tiuxetan; Radiation: yttrium Y 90 ibritumomab tiuxetan; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Drug: sirolimus — Given PO
  Other Names: AY 22989; Rapamune; rapamycin; SLM
Drug: tacrolimus — Given PO or IV
  Other Names: FK 506; Prograf
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo APBSCT
Radiation: indium In 111 ibritumomab tiuxetan — Given IV
  Other Names: IDEC-In2B8
Radiation: yttrium Y 90 ibritumomab tiuxetan — Given IV
  Other Names: 90Y ibritumomab tiuxetan; IDEC Y2B8; Y90 Zevalin; Y90-labeled ibritumomab tiuxetan
Other: laboratory biomarker analysis — Correlative Studies

SUMMARY:
RATIONALE: Giving monoclonal antibody therapy, radioimmunotherapy, and chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the stem cells from a related donor that do not exactly match the patient's blood, are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus and sirolimus before and after transplant may stop this from happening.

PURPOSE: This phase II trial is studying the side effects and how well giving indium In 111 ibritumomab tiuxetan and yttrium y 90 ibritumomab tiuxetan together with rituximab, fludarabine, melphalan, and donor stem cell transplant works in treating patients with B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To evaluate the safety and efficacy of a preparative regimen of Yttrium-90 (90^Y)- labeled anti-cluster of differentiation (CD)20 monoclonal antibody (MAb) (yttrium Y 90 ibritumomab tiuxetan) in combination with fludarabine (fludarabine phosphate) and melphalan followed by allogeneic hematopoietic stem cell transplant (APBSCT) for treatment of patients with B-cell low-grade non-Hodgkin lymphoma (LG NHL), intermediate-grade non-Hodgkin lymphoma (IG NHL) and mantle cell lymphoma (MCL). II. To evaluate the short- and long-term complications of this new preparative regimen, including rates of engraftment, acute and chronic graft-versus-host-disease (GVHD) and infectious complications. III. To estimate the disease response rate, disease relapse (progression) rate, and non-relapse mortality rate. IV. To perform exploratory studies that seek to measure/characterize the expression of costimulatory molecules and impact of these molecules on the natural killer (NK) and T cells of a subset of lymphoma patients pre- post- allogeneic stem cell transplant (ASCT) and the stem cell product from a portion of sibling donors.

OUTLINE: REDUCED-INTENSITY CONDITIONING: Patients receive rituximab intravenously (IV) followed by indium In-111 ibritumomab tiuxetan IV over 10 minutes on day -21 and rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day -14. Patients also receive fludarabine phosphate IV on days -9 to -5 and melphalan IV on day -4.

STEM CELL TRANSPLANTATION: Patients undergo APBSCT on day 0.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV or orally (PO) and sirolimus PO beginning on day -3 and continuing for up to 6 months with taper.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* 6/6/human leukocyte antigen (HLA) matched sibling donor or related donor, or acceptable matched unrelated donor
* Biopsy (Bx) proven diagnosis of LG (including small lymphocytic lymphoma [SLL]/chronic lymphocytic leukemia [CLL], lymphoplasmacytic lymphoma, marginal zone, mucosa-associated lymphoid tissue [MALT] lymphoma and follicular lymphoma [FL] grade 1 and 2), IG (FL grade 3 and DLCL) or MCL NHL
* Prior demonstrated monoclonal CD20+ malignant B-Cell population in lymph nodes and/or BM Bx specimen
* LG NHL; must have relapsed after achieving a complete response (CR) or partial response (PR) to prior therapy or have never responded to prior therapy, including chemotherapy and/or MAb therapy
* MCL NHL in any disease state
* Other aggressive B-cell lymphomas (excluding Burkitt lymphoma or Burkitt-like lymphoma) having had at least one relapse or having been refractory to chemotherapy
* Bone marrow (BM) aspiration and Bx ( =< 42 days prior to imaging dose) which show < 25% lymphomatous involvement of total cellularity; in CLL, peripheral lymphocyte count < 5000/mm^3
* Salvage chemotherapy/MAbs to reduce BM lymphomatous involvement and reduce disease bulk allowed
* Normal renal function test with serum creatinine of =< 1.5 mg/dl, or a creatinine clearance of >= 60 ml/min
* Adequate pulmonary function as measured by forced expiratory volume in one second (FEV1) > 65% of predicted measured, or a diffusing capacity of carbon monoxide (DLCO) >= 50% of predicted measured
* Cardiac Ejection fraction of > 50% by Echocardiogram (ECHO) or multi gated acquisition (MUGA)
* Adequate liver function tests with a bilirubin of =< 1.5 x normal and serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) =< 2 x normal
* Negative Human Immunodeficiency Virus (HIV) antibody
* Karnofsky Performance Status (KPS) > 80
* No active Central Nervous System (CNS) disease or prior history of CNS disease
* Involved field External Beam Therapy (EBT) to area excluding lung, heat, liver, and kidney allowed, but evaluated on a case-by-case basis
* Recovery from last therapy and therapy dose (Y-90 Zevalin) must be >= 4 weeks from prior systemic chemotherapy
* DONOR: Age < 75 years
* DONOR: HLA genotypically identical related donor or acceptable matched unrelated donor
* DONOR: Must consent to G-CSF administration and leukapheresis for matched sibling donor, but for unrelated donor, the donor will sign a standard consent for donation at their designated donor or collection center
* DONOR: Must have adequate veins for leukapheresis or agree to placement of a Central Venous Catheter (CVC [femoral, subclavian])

Exclusion Criteria:

* Presence of Human Anti-Zevalin Antibody (HAZA)
* Prior radioimmunotherapy (RIT)
* Prior AHSCT; but prior aHSCT is allowed; prior fractionated total body irradiation (FTBI) in the conditioning regimen will be evaluated on an individual basis
* Prior malignancy, except for: adequately treated basal cell or squamous cell skin cancer; adequately treated noninvasive carcinomas; or other cancer from which the patient has been disease-free for at least 5 years; myelodysplastic syndromes (MDS) is excluded from this criterion
* Active evidence of Hepatitis B or C infection; hepatitis B surface antigen positive
* Total peripheral lymphocyte count > 5,000/mm^3 if SLL/CLL
* Burkitt lymphoma or Burkitt-like lymphoma
* DONOR: Age < 12 years
* DONOR: Identical twin
* DONOR: Pregnancy
* DONOR: HIV infection
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to G-CSF
* DONOR: Current serious systemic illness or any disease that may preclude the use of G-CSF (eg, recent thromboembolic event); for unrelated donors, considered ineligible by National Marrow Donor Program (NMDP) donor evaluation center

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-10-03 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mei, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Mei M, Palmer J, Tsai NN, Simpson J, O'Hearn J, Stein A, Forman S, Spielberger R, Cai JL, Htut M, Nakamura R, Al Malki MM, Herrera A, Wong J, Nademanee A. Results of a Phase II Trial of Allogeneic Hematopoietic Stem Cell Transplantation Using 90Y-Ibritumomab Tiuxetan (Zevalin) in Combination With Fludarabine and Melphalan in Patients With High-Risk B-Cell Non-Hodgkin's Lymphoma. Clin Lymphoma Myeloma Leuk. 2023 Sep;23(9):e268-e276. doi: 10.1016/j.clml.2023.05.011. Epub 2023 May 23. PMID 37301631

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.4 mCi 90Y-Ibritumomab Tiuxetan: Patients receive rituximab IV followed by indium In-111 ibritumomab tiuxetan IV over 10 minutes on day -21 and rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day -14. Patients also receive fludarabine phosphate IV on days -9 to -5 and melphalan IV on day -4. Patients undergo APBSCT on day 0. GVHD PROPHYLAXIS: Patients receive tacrolimus IV or PO and sirolimus PO beginning on day -3 and continuing for up to 6 months with taper.
  rituximab: Given IV fludarabine phosphate: Given IV melphalan: Given IV sirolimus: Given PO tacrolimus: Given PO or IV allogeneic hematopoietic stem cell transplantation: Undergo APBSCT indium In 111 ibritumomab tiuxetan: Given IV yttrium Y 90 ibritumomab tiuxetan: Given IV
Period: Overall Study
Arm/Group | 0.4 mCi 90Y-Ibritumomab Tiuxetan
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 0.4 mCi 90Y-Ibritumomab Tiuxetan
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 55 [27 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 34
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Relapse/Progression Rate at Two Years
Description: The primary endpoint was 2-year cumulative incidence of relapse/progression (RP), defined as time from alloHCT to disease recurrence or progression. Cumulative incidences for RP was generated in a competing-risk setting, given that death events were competing events.
Time Frame: From the initial treatment to the last disease assessment, up to two years
Measure: Number (95% Confidence Interval); unit: percentage of cumulative incidence
Arm/Group | 0.4 mCi 90Y-Ibritumomab Tiuxetan
Number analyzed (Participants) | 41
percentage of cumulative incidence | 20 [10 to 36]

2. Secondary Outcome: Overall Survival at Two Years
Description: Overall survival (OS) was measured from initial treatment to death from any cause. It was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula.
Time Frame: From the initial treatment to the last disease assessment, up to two years
Measure: Number (95% Confidence Interval); unit: percentage of survival probability
Arm/Group | 0.4 mCi 90Y-Ibritumomab Tiuxetan
Number analyzed (Participants) | 41
percentage of survival probability | 63 [47 to 76]

3. Secondary Outcome: Progression-free Survival at Two Years
Description: Progression-free survival (PFS) was measured from initial treatment to disease progression or death from any cause, whichever came first. It was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula.
Time Frame: From the initial treatment to the last disease assessment, up to two years
Measure: Number (95% Confidence Interval); unit: percentage of survival probability
Arm/Group | 0.4 mCi 90Y-Ibritumomab Tiuxetan
Number analyzed (Participants) | 41
percentage of survival probability | 61 [44 to 74]

ADVERSE EVENTS:
Time Frame: From initial treatment to off study, up to 5 years.
Arm/Group | 0.4 mCi 90Y-Ibritumomab Tiuxetan
All-Cause Mortality (participants affected / at risk) | 24/41
Serious Adverse Events (participants affected / at risk) | 28/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.4 mCi 90Y-Ibritumomab Tiuxetan (N=41)
Chyle or lymph leakage (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, GI (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory (Blood and lymphatic system disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Blood and lymphatic system disorders) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 3 (4)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 2 (2)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 7 (9)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4)
Vomiting (Gastrointestinal disorders) | 2 (3)
Fever (General disorders) | 4 (4)
Pain (General disorders) | 3 (10)
Hepatobiliary/Pancreas - Other (Specify, __) (Hepatobiliary disorders) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Febrile neutropenia (Infections and infestations) | 2 (2)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 4 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 17 (34)
Infection, Bacterial (Infections and infestations) | 7 (8)
Infection, Fungal (Infections and infestations) | 1 (1)
Infection, Viral (Infections and infestations) | 3 (4)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 2 (2)
Viral hepatitis (Infections and infestations) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2 (2)
Acidosis (metabolic or respiratory) (Investigations) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
Amylase (Investigations) | 2 (2)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
Lipase (Investigations) | 2 (2)
Sodium, serum-low (hyponatremia) (Investigations) | 1 (1)
Secondary Malignancy - possibly related to cancer treatment (Specify, __) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (26)
Mood alteration (Nervous system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 2 (3)
Obstruction, GU (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.4 mCi 90Y-Ibritumomab Tiuxetan (N=41)
Bone marrow cellularity (Blood and lymphatic system disorders) | 14 (20)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1 (1)
Edema:head and neck (Blood and lymphatic system disorders) | 19 (21)
Edema:limb (Blood and lymphatic system disorders) | 35 (51)
Edema:trunk/genital (Blood and lymphatic system disorders) | 5 (5)
Haptoglobin (Blood and lymphatic system disorders) | 5 (5)
Hematoma (Blood and lymphatic system disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 41 (126)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 7 (9)
Hemorrhage, GI (Blood and lymphatic system disorders) | 22 (31)
Hemorrhage, GU (Blood and lymphatic system disorders) | 20 (24)
Hemorrhage, pulmonary/upper respiratory (Blood and lymphatic system disorders) | 20 (22)
Hemorrhage/Bleeding - Other (Specify, __) (Blood and lymphatic system disorders) | 3 (3)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 3 (3)
Iron overload (Blood and lymphatic system disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 41 (114)
Lymphatics - Other (Specify, __) (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 41 (143)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 41 (142)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 6 (7)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 14 (15)
Phlebitis (including superficial thrombosis) (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 41 (103)
Thrombosis/embolism (vascular access-related) (Blood and lymphatic system disorders) | 3 (3)
Thrombosis/thrombus/embolism (Blood and lymphatic system disorders) | 2 (2)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 10 (12)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 3 (3)
Conduction abnormality/atrioventricular heart block (Cardiac disorders) | 1 (3)
Hypertension (Cardiac disorders) | 30 (79)
Hypotension (Cardiac disorders) | 16 (19)
Left ventricular diastolic dysfunction (Cardiac disorders) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 6 (7)
Palpitations (Cardiac disorders) | 2 (2)
Pericardial effusion (non-malignant) (Cardiac disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Prolonged QTc interval (Cardiac disorders) | 11 (15)
Pulmonary hypertension (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 30 (59)
Ventricular arrhythmia (Cardiac disorders) | 2 (2)
Hearing (Ear and labyrinth disorders) | 2 (4)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Cushingoid appearance (Endocrine disorders) | 10 (11)
Hot flashes/flushes (Endocrine disorders) | 2 (2)
Neuroendocrine:ADH secretion abnormality (e.g., SIADH or low ADH) (Endocrine disorders) | 2 (3)
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 1 (1)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Dry eye syndrome (Eye disorders) | 6 (7)
Glaucoma (Eye disorders) | 1 (2)
Nystagmus (Eye disorders) | 1 (1)
Ocular surface disease (Eye disorders) | 2 (2)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 2 (3)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 2 (2)
Proptosis/enophthalmos (Eye disorders) | 1 (3)
Vision-blurred vision (Eye disorders) | 4 (4)
Watery eye (epiphora, tearing) (Eye disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 35 (51)
Ascites (non-malignant) (Gastrointestinal disorders) | 6 (8)
Colitis (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 18 (19)
Dehydration (Gastrointestinal disorders) | 11 (11)
Dental: teeth (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 41 (78)
Distension/bloating, abdominal (Gastrointestinal disorders) | 21 (26)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 31 (32)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 7 (8)
Esophagitis (Gastrointestinal disorders) | 6 (6)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 10 (10)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 6 (6)
Heartburn/dyspepsia (Gastrointestinal disorders) | 21 (28)
Hemorrhoids (Gastrointestinal disorders) | 10 (11)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 5 (5)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 40 (75)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 36 (57)
Nausea (Gastrointestinal disorders) | 41 (61)
Proctitis (Gastrointestinal disorders) | 2 (2)
Salivary gland changes/saliva (Gastrointestinal disorders) | 3 (3)
Stricture/stenosis (including anastomotic), GI (Gastrointestinal disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 9 (11)
Ulcer, GI (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 37 (45)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 41 (93)
Fever (General disorders) | 14 (15)
Insomnia (General disorders) | 31 (39)
Pain (General disorders) | 40 (463)
Pain - Other (Specify, __) (General disorders) | 15 (21)
Rigors/chills (General disorders) | 28 (32)
Sweating (diaphoresis) (General disorders) | 9 (10)
Weight gain (General disorders) | 25 (26)
Weight loss (General disorders) | 31 (64)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 2 (2)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3 (3)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2)
Autoimmune reaction (Immune system disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 10 (13)
Febrile neutropenia (Infections and infestations) | 26 (26)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 20 (30)
Infection - Other (Specify, __) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 29 (77)
Infection with unknown ANC (Infections and infestations) | 4 (4)
Infection, Bacterial (Infections and infestations) | 15 (27)
Infection, Fungal (Infections and infestations) | 3 (3)
Infection, Viral (Infections and infestations) | 15 (21)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 1 (4)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 35 (65)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 38 (71)
Acidosis (metabolic or respiratory) (Investigations) | 3 (3)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 40 (71)
Alkaline phosphatase (Investigations) | 23 (44)
Alkalosis (metabolic or respiratory) (Investigations) | 1 (1)
Amylase (Investigations) | 2 (3)
Bicarbonate, serum-low (Investigations) | 29 (39)
Bilirubin (hyperbilirubinemia) (Investigations) | 15 (18)
CPK (creatine phosphokinase) (Investigations) | 1 (1)
Calcium, serum-high (hypercalcemia) (Investigations) | 9 (10)
Calcium, serum-low (hypocalcemia) (Investigations) | 36 (50)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 28 (48)
Creatinine (Investigations) | 24 (36)
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 3 (5)
Glucose, serum-high (hyperglycemia) (Investigations) | 39 (85)
Glucose, serum-low (hypoglycemia) (Investigations) | 16 (20)
Hemoglobinuria (Investigations) | 1 (1)
Lipase (Investigations) | 1 (2)
Magnesium, serum-high (hypermagnesemia) (Investigations) | 10 (11)
Magnesium, serum-low (hypomagnesemia) (Investigations) | 40 (63)
Phosphate, serum-low (hypophosphatemia) (Investigations) | 30 (52)
Potassium, serum-high (hyperkalemia) (Investigations) | 13 (15)
Potassium, serum-low (hypokalemia) (Investigations) | 39 (73)
Proteinuria (Investigations) | 10 (11)
Sodium, serum-high (hypernatremia) (Investigations) | 1 (1)
Sodium, serum-low (hyponatremia) (Investigations) | 38 (74)
Triglyceride, serum-high (hypertriglyceridemia) (Investigations) | 39 (86)
Uric acid, serum-high (hyperuricemia) (Investigations) | 6 (7)
Obesity (Metabolism and nutrition disorders) | 30 (126)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 3 (5)
Joint-effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 37 (79)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Secondary Malignancy - possibly related to cancer treatment (Specify, __) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (7)
Cognitive disturbance (Nervous system disorders) | 3 (3)
Confusion (Nervous system disorders) | 7 (9)
Dizziness (Nervous system disorders) | 20 (26)
Encephalopathy (Nervous system disorders) | 2 (2)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 8 (9)
Mental status (Nervous system disorders) | 1 (1)
Mood alteration (Nervous system disorders) | 31 (80)
Neurology - Other (Specify, __) (Nervous system disorders) | 3 (3)
Neuropathy: cranial (Nervous system disorders) | 2 (6)
Neuropathy: motor (Nervous system disorders) | 3 (4)
Neuropathy: sensory (Nervous system disorders) | 22 (26)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 4 (4)
Seizure (Nervous system disorders) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 8 (9)
Syncope (fainting) (Nervous system disorders) | 4 (4)
Tremor (Nervous system disorders) | 10 (10)
Bladder spasms (Renal and urinary disorders) | 3 (3)
Cystitis (Renal and urinary disorders) | 4 (4)
Incontinence, urinary (Renal and urinary disorders) | 3 (3)
Obstruction, GU (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 8 (9)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 4 (4)
Urine color change (Renal and urinary disorders) | 4 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Libido (Reproductive system and breast disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 19 (24)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 30 (35)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (31)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 20 (34)
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 2 (2)
FEV(1) (Respiratory, thoracic and mediastinal disorders) | 13 (16)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (17)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 20 (27)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 17 (25)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 24 (36)
Vital capacity (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Syndromes - Other (Specify, __) (Investigations) | 13 (13)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 18 (20)
Burn (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 7 (11)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (17)
Flushing (Skin and subcutaneous tissue disorders) | 16 (18)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 23 (33)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 (14)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 1 (2)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 17 (21)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 39 (60)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 8 (11)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT00577278/Prot_SAP_000.pdf